CLINICAL TRIAL: NCT01574820
Title: Role of Rosiglitazone Treatment and Secondary Prevention of Cardiovascular Events in Patients With Pre-Diabetes Mellitus and Coronary Artery Disease
Brief Title: Role of Rosiglitazone on Pre-Diabetes Mellitus and Coronary Artery Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCKUH HR95-10
Record Dates: First submitted 2012-04-04; First posted 2012-04-10 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Prediabetes; Coronary Artery Disease; Insulin Resistance; Glucose Intolerance
Keywords: prediabetes; coronary artery disease; insulin resistance; glucose intolerance
MeSH Terms: conditions — Prediabetic State; Coronary Artery Disease; Insulin Resistance; Glucose Intolerance | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo tablet
- rosiglitazone (4 mg)/day (Experimental)
  Interventions: Drug: rosiglitazone (4 mg)/day

INTERVENTIONS:
Drug: placebo tablet — placebo tablet for 6 months
  Arms: placebo
Drug: rosiglitazone (4 mg)/day — rosiglitazone (4 mg)/day for 6 months
  Arms: rosiglitazone (4 mg)/day

SUMMARY:
Objectives:

The investigators examined whether rosiglitazone, a thiazolidinedione (TZD), is beneficial for pre-diabetes mellitus (DM) adults with documented coronary artery disease (CAD).

Background:

Microvascular and macrovascular complications are common in type 2 DM. There is no evidence about the effects of TZDs, synthetic peroxisome proliferator-activated receptor (PPAR)-γ activators (insulin sensitizers and adipose transcriptional regulation and anti-inflammatory process activators) on pre-DM patients with documented CAD.

DETAILED DESCRIPTION:
Materials and Methods:

This is a randomized, double-blind, placebo-controlled study, patients will be randomly assigned to the TZD group and to the placebo group with a 6-month treatment period.

Biomarkers will also examined before and 6 months post-treatment during the trial.

The primary end-points will be the diagnosis of major cardiovascular events: myocardial infarction, overt heart failure, and surgery or coronary intervention for CAD.

ELIGIBILITY:
Inclusion Criteria:

* documented CAD by angiography
* insulin resistance or glucose intolerance
* 18 to 80 years of age

Exclusion Criteria:

* under DM treatment
* allergy to TZD
* active inflammation
* chronic disease under NSAID treatment
* active heart failure
* unwilling or unable to sign inform consents

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2006-11; Primary Completion 2010-08 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
major cardiovascular events, including myocardial infarction, overt heart failure, and surgery or coronary intervention for CAD | at least 6 months follow-up of MACEs
  Primary end points: The primary end-point was defined as major cardiovascular events, including myocardial infarction, overt heart failure, and surgery or coronary intervention for CAD.

SECONDARY OUTCOMES:
Biomarkers measurements | Biomarkers were taken before the trial and 6 months later
  Resistin and adiponectin will be measured to evaluate insulin resistance; CCL/MCP-1 and hsCRP were also analyzed to evaluate inflammation status changes.
  Several vascular associated remodeling markers and proteins will also be measured.